CLINICAL TRIAL: NCT06872567
Title: Resorbable Embolization MicroSpheres for OsteoaRthritis Benefit
Brief Title: Randomized Controlled Study Evaluating Genicular Artery Embolization Against Intra-Articular Corticosteroid Knee Injection for Osteoarthritic Knee Pain
Acronym: RESORB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: North American Science Associates Ltd. (Network)
Collaborators: Next Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: US037031
Record Dates: First submitted 2025-02-27; First posted 2025-03-12 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis (Knee OA)
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Control (Active Comparator)
  Interventions: Drug: Corticosteroid Injection
- Device: GAE (Experimental)
  Interventions: Device: genicular artery embolization

INTERVENTIONS:
Device: genicular artery embolization — genicular artery embolization
  Arms: Device: GAE
Drug: Corticosteroid Injection — Corticosteroid Injection
  Arms: Control

SUMMARY:
Multi-center, prospective, randomized trial of GAE using Nexsphere-F against steroid injection

ELIGIBILITY:
Inclusion Criteria:

* Patient has localized knee pain
* Must be an appropriate candidate for arterial vascular access procedure

Exclusion Criteria:

* Known sensitivity or allergy to implant materials
* Unable or unwilling to comply with study requirements

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 and 12-month post treatment
  Changes in total Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score. Scale ranges from 0 to 96 with higher scores equating to greater pain, stiffness and difficulty with activities of daily living.
Serious Adverse Events (SAE) | Treatment, 1,3,6,9 and 12-month post treatment

SECONDARY OUTCOMES:
WOMAC total score | 9 month post treatment
  Changes in total Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score. Scale ranges from 0 to 96 with higher scores equating to greater pain, stiffness and difficulty with activities of daily living

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided